CLINICAL TRIAL: NCT02285946
Title: Alveolar Recruitment Maneuvers: Comparison of Supine to Prone Position During Major Spinal Surgery
Brief Title: Comparison of Supine to Prone Position During Major Spinal Surgery
Acronym: MRA-RACHIS
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6032
Record Dates: First submitted 2014-10-02; First posted 2014-11-07 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Osteotomies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: major spine surgery

SUMMARY:
During mechanical ventilation, the alveolar recruitment maneuver (ARM) is to apply a positive end-expiratory pressure (PEEP) (generally 30 cm H2O) for a period of at least 30 seconds. The realization of MRA is one of three main elements of mechanical ventilation called "protective". This ventilatory strategy, originally described for the ventilation of acute respiratory distress syndrome (ARDS), and pulmonary and during abdominal surgery is based on a decrease tidal volumes, optimization of PEEP and the realization of MRA. Protective ventilation limit the occurrence of atelectasis, the surdistentions and, ultimately, significantly decreases postoperative complications.

The MRA is currently recommended in the "major" surgery. Most spine surgery (eg transpedicular fixation) used in this definition, the MRA are indicated and now commonly used. This type of surgery requires further positioning the patient in the prone position (DV). The DV modifies the compliance of the chest respiratory characteristics and changes (increase in insufflation pressure) and hemodynamic (decreased venous return) of the patient.

Respiratory and haemodynamic effects of MRA made VIS at major spine surgery are not known. The aim of this observational study, non-interventional, is to compare the hemodynamic and respiratory effects of MRA performed in DV to those of MRA performed in the prone position (DD).

The investigators hypothesis is that the respiratory and hemodynamic consequences of MRA performed in DV is different from those conducted in DD. A better understanding of hemodynamic and respiratory characteristics of MRA performed in DV would provide a more tailored to this type of surgery respiratory optimization strategy and reduce respiratory complications of this surgery.

ELIGIBILITY:
Inclusion Criteria:

Adult patient

Patient operated major spine surgery, including:

* The transpedicular osteotomies
* Tumor spinal surgery (sarcoma, osteosarcoma) or metastatic
* Degenerative spinal surgery on multiple vertebral levels and degraded land
* Surgery of scoliosis

Exclusion Criteria:

* Inability to give informed patient information (eg difficulty of understanding)
* Patient under guardianship - Patient pregnant or during lactation - Detainees or under judicial protection.
* contraindications to MRA: emphysema, pneumothorax, major hypovolemia, hemodynamic instability defined as systolic blood pressure below 90 mmHg or tachycardia greater than 110 bpm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient operated major spine surgery, including:
  * The transpedicular osteotomies
  * Tumor spinal surgery (sarcoma, osteosarcoma) or metastatic
  * Degenerative spinal surgery on multiple vertebral levels and degraded land
  * Surgery of scoliosis
  * Recovery of spinal surgery on several levels
  * Sepsis spinal presumed origin
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
The hemodynamic and respiratory data are collected before, during and after the completion of 3 ARM (alveolar recruitment maneuver): | T1: ARM (in a supine position) (before setting prone position); T2: ARM (prone position) ; T3: ARM at acute respiratory distress syndrome [ARDS] (end of intervention, after supine position); (* At the end of ARM, only hemodynamic data are collected)

CONTACTS AND LOCATIONS:
Overall Officials: COLLANGE Olivier, MD, Principal Investigator — Strasbourg University Hospital, France
Locations (1):
- Service D'Anesthesiologie - Nhc, Strasbourg, France